CLINICAL TRIAL: NCT06578234
Title: Hyperemic mYocardial Perfusion by adEnosine at diffeRent Doses
Acronym: HYPER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2023-505248-20-00
Record Dates: First submitted 2024-08-15; First posted 2024-08-29 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Chronic Coronary Syndrome; Coronary Artery Disease; Ischemic Heart Disease
Keywords: Myocardial perfusion; Cardiac Magnetic Resonance; Adenosine
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia | interventions — Adenosine

STUDY DESIGN:
Intervention Model Description: The subjects will be randomized to start with one of the two adenosine doses, followed by the other dose 10 minutes later during the same examination.
Who Masked: Participant
Masking Description: The subject will be blinded to the order of adenosine doses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Start standard dose adenosine followed by high dose adenosine (Active Comparator): Subjects randomized to this arm will undergo the first stress perfusion acquisition with a dose of 140 μg/kg/min adenosine, followed by a second stress perfusion acquisition with the dose of 210 μg/kg/min adenosine.
  Interventions: Drug: Adenosine
- Start high dose adenosine followed by standard dose adenosine (Active Comparator): Subjects randomized to this arm will undergo the first stress perfusion acquisition with a dose of 210 μg/kg/min adenosine, followed by a second stress perfusion acquisition with the dose of 140 μg/kg/min adenosine.
  Interventions: Drug: Adenosine

INTERVENTIONS:
Drug: Adenosine — Standard dose 140 μg/kg/min and high dose 210 μg/kg/min adenosine

SUMMARY:
Adenosine is a commonly used pharmaceutical stressor at cardiac magnetic resonance examinations to assess suspected chronic coronary syndrome (CCS). However, several studies have reported that the current use of adenosine does not induce adequate hyperemic response in a substantial number of patients, leading to false diagnostics. The aim of this trial is to investigate the hyperemic effect of the standard dose of adenosine (140 microgram/kg/min) to the high dose of adenosine (210 microgram/kg/min) to improve the diagnostic methods using adenosine as a stressor and ultimately improve treatment decisions and patient prognosis in CCS.

ELIGIBILITY:
Inclusion Criteria:

Patients:

1. The subject has given their written consent to participate in the trial.
2. Are referred to Department of Clinical Physiology, Skåne University Hospital, for suspected or known CCS or heart failure
3. Matches the inclusion criteria for sex and age (6 females and 6 males from each group in each age decade from 40 to >80 years old)
4. Matches the inclusion criteria for no known heart failure (group b) or known heart failure (group c)
5. No caffein intake <24h prior to the examination

Healthy volunteers:

1. The subject has given their written consent to participate in the trial.
2. Matches the inclusion criteria for sex and age (6 females and 6 males from each group in each age decade from 40 to >80 years old)
3. No caffein intake <24h prior to the examination

Exclusion Criteria:

Patients:

1. Acute referral (in-house patients)
2. Clinically unstable
3. Acute chest pain
4. Severe or decompensated heart failure
5. Non sinus rhythm (e.g. atrial fibrillation)
6. Asthma or severe chronic obstructive pulmonary disease
7. Known chronic renal failure (eGFR <45mL/min/1.73m2)
8. AV-block II or III
9. Left Bundle Branch Block
10. Systolic blood pressure <90 mmHg or >230 mmHg at rest
11. Increased intracranial pressure
12. Known allergy or adverse reaction to adenosine or mannitol
13. Known allergy or adverse reaction to gadolinium contrast agents
14. Treatment with medication containing dipyradimol or teofyllamin/teofyllin
15. Claustrophobia
16. Devices contraindicated to CMR imaging (pacemaker, implants, intracranial clips etc)
17. Pregnancy or breast feeding (screened by question only)
18. Inability to give informed consent due to mental state, language difficulties etc

Healthy volunteers:

1. Any of the exclusion criteria for patients
2. Blood pressure > 140/90 measured according to clinical routine
3. Known systemic disease
4. Known cardiac disease
5. Cardiovascular medication
6. Medication that might influence cardiovascular health
7. Smoking

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial hyperemia | During adenosine infusion, 4-6 minutes
  The primary outcome measure is assessed by quantitative myocardial perfusion CMR imaging (ml/min/g).

SECONDARY OUTCOMES:
Heart rate response | During adenosine infusion, 4-6 minutes
  Compare heart rate (beat/min) at standard and high dose adenosine
Blood pressure response | During adenosine infusion, 4-6 minutes
  Compare systolic blood pressure (mmHg) at standard and high dose adenosine
Symptoms | During adenosine infusion, 4-6 minutes
  Compare presence of symptoms (evaluated using a Borg10-scale) at standard and high dose adenosine

OTHER OUTCOMES:
Sex | In questionnaire obtained approximately 30 minutes before CMR examination
  The association between sex (female and male) and adenosine response
Age | In questionnaire obtained approximately 30 minutes before CMR examination
  The association between age (years) and adenosine response
Ejection fraction | Measured in the obtained short-axis cine images within approximately 6 months after acquisition
  The association between ejection fraction (%) assessed from CMR images and adenosine response
Serum-caffeine | Blood samples are analysed within 9 months
  The association between serum caffeine levels (mg/L) assessed from blood samples and adenosine response

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Physiology, Department of Clinical Sciences Lund, Lund University, Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No